CLINICAL TRIAL: NCT05031572
Title: New Energy-sensing Metabolites: Beneficial Effects on Metabolic Health in Obesity Comparing Diary Caloric Restriction vs Intermittent Fasting. A Randomized Cross-over Study
Brief Title: Energy -Sensing Metabolites in Caloric Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Joan Josep Vendrell, professor, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PI20/00338
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Insulin Sensitivity/Resistance; Diabetes Type 2
Keywords: obesity; diabetes; intermittent fasting; energy-sensing metabolites
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2; Diabetes Mellitus; Intermittent Fasting | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: clinical study: randomized, cross-over design, study participants will consume either lifestyle recommendations for a healthy Mediterranean diet under a continued caloric restriction diet (DCR) or will undertake an intermittent (IF) protocol
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional caloric restriction diet (Other): (DCR protocol): lifestyle recommendations for a healthy Mediterranean diet under a continued daily caloric restriction diet
  Interventions: Other: dietary intervention
- Intermitent fasting (Other): Fasting for two days (non-consecutive) out of seven, with the fasting days separated by at least one day.
  Interventions: Other: dietary intervention

INTERVENTIONS:
Other: dietary intervention — Chronic caloric restriction diet vs intermittent fasting on energy sensing metabolites and metabolic homeostasis

SUMMARY:
General integrated goal of the coordinated project:

To elucidate the role of succinate and other metabolites derived from the intestinal microbiota such as Short Chain Fatty Acids (SCFAs), as energy sensing metabolites in the context of obesity and type 2 diabetes (T2D).

Specific objectives of Subproject 1 (SP1): 1a. - To investigate whether intermittent fasting (IF) is better than Continued Daily Caloric Restriction (DCR) in terms of metabolic improvement through the study of: 1) the dynamics of gastrointestinal hormones and energy sensing metabolites, 2) the intestinal microbiome, 3) variability on succinate and SCFAs, MCFAs and Biliary Acid after weight loss; Methodology: clinical study: randomized, cross-over design, study participants (n=15) will consume either lifestyle recommendations for a healthy Mediterranean diet under a continued caloric restriction diet (DCR) or will undertake an intermittent (IF) protocol. Clinical, anthropometrical and functional studies. Metabolomics for gut derived metabolites in plasma. Enteroendocrine gastrointestinal dynamics. Metagenomic analysis.

DETAILED DESCRIPTION:
To investigate whether IF is better than DCR in terms of metabolic improvement through the study of:

1. the dynamics of gastrointestinal hormones and energy sensing metabolites
2. the intestinal microbiome
3. variability on succinate and SCFAs MCFAs and BA after weight loss

Human study protocol:

A pilot clinical trial in human study participants will be assayed. Participants for intermittent fasting (IF) will be asked to fast for 24 hours on two days of the week (2/5 protocol).

1A.-Design: Utilizing a randomized, cross-over design, study participants (n=15) will consume either lifestyle recommendations for a healthy Mediterranean diet under a continued daily caloric restriction diet (DCR) or will undertake an intermittent (IF) protocol. Each study period will be 8 weeks - total study period will be 16 weeks + a 4-week washout period between dietary exposures. The study participants will be adults who have obesity with a Body Mass Index (BMI)25 kg/m2 and 40 kg/m2 and have no contraindications for intermittent fasting (see inclusion and exclusion criteria below).

ELIGIBILITY:
Inclusion Criteria:

* White men and women between 18 and 65 years of age.
* BMI range between 25 and 40 kg/m2
* Absence of underlying pathology in medical and physical examination, except for those related to excess weight.
* Signature of the informed consent for participation in the study.

Exclusion Criteria:

* Serious systemic disease not related to obesity, such as cancer, kidney or severe liver disease.
* Systemic diseases with intrinsic inflammatory activity (autoimmune diseases such as rheumatoid arthritis and asthma)
* Pregnancy and lactation.
* Vegetarians or subjects subjected to an irregular diet.
* Patients with severe eating disorders.
* Patients with clinical symptoms and signs of infection in the previous month.
* Patients with chronic anti-inflammatory steroid treatments and/or nonsteroidal anti-inflammatory drugs.
* Recent antibiotic treatment.
* Psychiatric history.
* Uncontrolled alcoholism or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
To investigate whether IF is better than DCR in terms of metabolic improvement through the study (change in the secretory pattern of glucose) | basal and after 8 weeks
  Plasma concentrations of glucose during a meal test
To investigate whether IF is better than DCR in terms of metabolic improvement through the study (change in the secretory pattern of insulin) | basal and after 8 weeks
  Plasma concentrations of insulin during a meal test
To investigate whether IF is better than DCR in terms of metabolic improvement through the study (change in the secretory pattern of glucose after crossing arm) | at beginning of week 12 vs week 20
  Plasma concentrations of glucose during a meal test
To investigate whether IF is better than DCR in terms of metabolic improvement through the study (change in the secretory pattern of insulin after crossing arm) | at beginning of week 12 vs week 20
  Plasma concentrations of insulin during a meal test

SECONDARY OUTCOMES:
1) the dynamics of gastrointestinal hormones and energy sensing metabolites | 8 weeks - 20 weeks
  GLP-1; GLP-2 during a meal test
2) Analysis of microbial species in fecal samples (gut flora) | 8 weeks - 20 weeks
  intestinal microbiome after each interventional period
variability on succinate after weight loss | 8 weeks - 20 weeks
  quantification of succinate
variability on Short-chain fatty acids (SCFAs) after weight loss | 8 weeks - 20 weeks
  quantification of SCFAs
variability on Medium-chain fatty acids (MCFAs) after weight loss | 8 weeks - 20 weeks
  quantification of MACFAs
variability on biliary acids (BA) after weight loss | 8 weeks - 20 weeks
  quantification of BA

CONTACTS AND LOCATIONS:
Overall Officials: Joan J Vendrell, PhD, Study Director — Director
Locations (1):
- Hospital Universitari Joan XXIII de Tarragona. IISPV, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No
Data sharing will be upon request directly to the PI

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT05031572/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT05031572/ICF_001.pdf